CLINICAL TRIAL: NCT04754854
Title: Reduction of Blood Recirculation in Veno-Venous ECMO Through Ultrasound Dilution Measurements (ECMO Circulation Study)
Brief Title: Reduction of Blood Recirculation in Veno-Venous ECMO
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Steffen Weber-Carstens, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA115620
Record Dates: First submitted 2020-09-14; First posted 2021-02-15 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Extracorporeal Membrane Oxygenation; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood which recirculates through the circuit of a veno-venous Extracorporeal Membrane Oxygenation (V-V ECMO) does not contribute to the systemic oxygenation of a patient on V-V ECMO and is called the recirculation fraction (Rf). Theoretically, the optimization of ECMO blood flow is possible using Rf measurements.

A prospective, observational study will be performed measuring the Rf of total ECMO blood flow in patients with acute respiratory distress syndrome (ARDS) on V-V ECMO with an ultrasound dilution technique.

ECMO blood flow will be optimized by reducing ECMO blood flow in accordance with the measured Rf as long as systemic oxygenation is not compromised.

DETAILED DESCRIPTION:
Based on data from the 'Blood Recirculation and vvECMO' trial (ClinicalTrials.gov ID: NCT03200314) (i.e. an expected frequency of successful blood flow reduction of 66.7%), using a one-sample Chi square test, a two-sided type-1 error of 5%, a power of 80%, a total of 68 patients is needed to show that the proportion of patients with a secure ECMO blood flow reduction is greater than 50%. Presumably, 136 Patients have to be included into the trial to study 68 patients with a relevant Rf since not all patients on V-V ECMO suffer from a high Rf.

ELIGIBILITY:
Patients aged 18 years or older requiring veno-venous ECMO for treatment of refractory hypoxemia in ARDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * patients aged 18 years or older
  * ARDS
  * veno-venous ECMO
  Exclusion Criteria:
  * age < 18 years
  * hemodynamic instability during measurement of recirculation
  * pregnancy
  * inability to obtain patient's consent or consent of legal guardian
Sampling Method: Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Successful ECMO blood flow reduction | Once within the first week after initiation of ECMO therapy
  Number of patients with a relevant recirculation fraction and successful ECMO blood flow reduction

SECONDARY OUTCOMES:
Recirculation fraction | Once within the first week after initiation of ECMO therapy
  Fraction of blood recirculating through the ECMO circuit
Arterial blood oxygen content | Once within the first week after initiation of ECMO therapy
  Arterial blood oxygen content before vs. after reduction of ECMO blood flow
Extracorporeal blood Flow | Once within the first week after initiation of ECMO therapy
  ECMO Blood Flow before vs. after reduction of ECMO blood flow
Extracorporeal gas flow | Once within the first week after initiation of ECMO therapy
  ECMO Sweep Gas flow
Length of ECMO therapy | Daily until the end of ECMO therapy (approximately 14 days)
  Days on ECMO
Cannula position and distance | Once within the first week after initiation of ECMO therapy
  The distance between the tip of drainage and return cannula will be measured in the existing medical imaging (e.g. CT scans)
Right heart dysfunction | Once within the first week after initiation of ECMO therapy
  Existing echocardiography will be evaluated for possible right heart dysfunction
Length of mechanical ventilation | Entire duration of the ICU stay (approximately 28 days)
  Length of mechanical ventilation
Complications of ECMO therapy | Length of ECMO therapy (approximately 14 days)
  Incidence of cannula or system changes (i.e. due to circuit clotting), complications attributed to ECMO therapy like bleeding complications from the cannulation site, transfusion requirements, hemolysis
ICU mortality | Entire duration of the ICU stay (approximately 28 days)
  ICU mortality
ICU length of stay | Entire duration of the ICU stay (approximately 28 days)
  ICU length of stay
Incidence of ICU-acquired organ dysfunctions and complications | Entire duration of the ICU stay (approximately 28 days)
  Cerebral-, cardiovascular-, cardiac- pulmonary-, gastrointestinal- and renal dysfunctions, ICU-acquired infections
ECMO blood flow over time | Daily until the end of ECMO therapy (approximately 14 days)
  ECMO blood and sweep gas flow over time
ECMO sweep gas flow over time | Daily until the end of ECMO therapy (approximately 14 days)
  ECMO sweep gas flow over time
Mobility at ICU discharge | Discharge from the ICU (approximately 28 days)
  Level of mobility the patient has reached at ICU discharge (recumbent, sitting, standing, walking with help, walking independently)
Weaning level at ICU discharge | Discharge from the ICU (approximately 28 days)
  Level of weaning reached at ICU discharge
Status of mechanical ventilation at ICU discharge | Discharge from the ICU (approximately 28 days)
  Status of mechanical ventilation at ICU discharge including all relevant settings and parameters
Level of organ dysfunction at ICU discharge | Discharge from the ICU (approximately 28 days)
  Sepsis-related Organ Failure Assessment Score at ICU discharge
Level of consciousness at ICU discharge | Discharge from the ICU (approximately 28 days)
  Glasgow Coma Scale at ICU discharge
Level of disease severity | Discharge from the ICU (approximately 28 days)
  Acute Physiology And Chronic Health Evaluation at ICU discharge
Hospital acquired infections related to ECMO therapy | Entire duration of ECMO therapy
  Infection/colonisation of the ECMO circuit
Bleeding and thrombembolic complications of ECMO therapy | Entire duration of ECMO therapy
  Bleeding complications, thrombembolic events, overall use of blood products and coagulation factors, electron microscopic evaluation of selected membranes after change or weaning of the ECMO circuit

CONTACTS AND LOCATIONS:
Overall Officials: Martin Russ, Dr. med., Principal Investigator — Charite University Hospital Berlin; Philipp A Pickerodt, Dr. med., Principal Investigator — Charite University Hospital Berlin; Vladimir Skrypnikov, Dr. med., Principal Investigator — Charite University Hospital Berlin; Steffen Weber-Carstens, Prof. Dr. med., Principal Investigator — Charite University Hospital Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No